CLINICAL TRIAL: NCT04344548
Title: Phase I / II Clinical Study of Immunotherapy Based on Adoptive Cell Transfer as a Therapeutic Alternative for Patients With COVID-19 in Colombia
Brief Title: Adoptive Cell Transfer for the Immunotherapy of COVID-19 in Colombia
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: The study did not get financed. Never get started.
Sponsor: Universidad Nacional de Colombia (Other)
Collaborators: Fundación Salud de los Andes (Other)
Responsible Party: Principal Investigator, Carlos Alberto Parra Lopez, Professor, Universidad Nacional de Colombia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UNAL FSA COVID; Estudio Clinico (Other: Fundación Salud de los Andes-Universidad Nacional)
Record Dates: First submitted 2020-04-10; First posted 2020-04-14 (Actual); Last update posted 2021-05-05 (Actual); Status verified 2021-04

CONDITIONS: COVID

STUDY DESIGN:
Intervention Model Description: Phase I/II immunotherapy with NK cells for mild infected COVID-19 patients
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment group (Experimental): Adult patients with COVID-19 infection with NEWS 2 score >4
  Interventions: Biological: Allogeneic NK transfer

INTERVENTIONS:
Biological: Allogeneic NK transfer — Three doses of allogeneic NK cell transfer

SUMMARY:
Immunotherapy based on Adoptive Cellular Transfer (ACT) uses several types of immune cells, including dendritic cells, cytotoxic T lymphocytes, lymphokine-activated killer cells, and NK cells. NK cell-based immunotherapies are an attractive approach for treating diseases because of their characteristic recognition and killing mechanisms; they are involved in the early defense against infectious pathogens and against MHC class-I-negative or -low-expressing targets without the requirement for prior immune sensitization of the host and are able to lyse target through the release of perforin and granzymes and using antibody-dependent cellular cytotoxicity pathways mediated by Fc receptor for IgG (CD16).

The aim of this project is to evaluate the safety and immunogenicity of allogeneic NK cells from peripheral blood mononuclear cells (PBMCs) of healthy donors in patients infected with COVID-19 collected by apheresis. This allows us to collect cGMP PBMCs and immunomagnetic remove several types of undesirable cells including B, T and CD33+ cells with enrichment of NK cells that will be expanded in bioreactors with GMP culture media (AIM-V) supplemented with human AB serum and GMP grade IL-2, and IL-15. After quality control verification the final NK cell product will be resuspended in 300 mL saline solution for intravenous infusion. Initially, we will enroll in this study ten COVID-19 infected adult patients with moderate symptoms (NEWS 2 scale score>4). Consent forms will be signed by the patient before the therapy. Patients will be treated with three different infusions of NK cells 48 h apart with 1, 10, and 20 million cells/kg body weight. We will follow the patients for any adverse effect, clinical response and immune effects by flow cytometry including markers for NK cells expressing different markers (CD158b, NKG2A, and IFN-y). We anticipated that the release of IFN-y by exogenous NK cells could attract other immune cell populations to boost the immune response against COVID-19.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years at the time of the evaluation
* Able and willing to understand the study, follow all study procedures, and provide written informed consent.
* Initial diagnosis of COVID-19 disease as defined by a molecular diagnostic test approved by the National Institute of Health positive for SARS-CoV-2
* Clinical presentation of moderate or severe (identified at the time of admission to the room by the National Early Warning Score NEWS-2; moderate >4)

Exclusion Criteria:

* Patients who are hospitalized for inpatient treatment or are currently being evaluated for possible hospitalization at the time of informed consent initiation.
* Oxygen saturation in ambient air of <92%
* History of Chronic Obstructive Pulmonary Disease (COPD)
* Participation in a clinical trial with or use of any investigational agent within 30 days prior to detection, or treatment with interferons (IFN) or immunomodulators within 12 months prior to detection
* Pregnant or lactating female patients.
* Current or previous history of decompensated liver disease (Child-Pugh Class B or C) or hepatocellular carcinoma
* Co-infected with the human immunodeficiency virus (HIV) or the hepatitis C virus (HCV)
* Significant abnormal laboratory test results on screening.
* Significant concurrent diseases and other comorbidities that may require intervention during the study.
* Concurrent use of any of the following medications: Therapy with an immunomodulatory agent. Current use of heparin o Coumadin. Received blood products within 30 days prior to study randomization. Use of hematological growth factors within 30 days prior to the randomization of the study. Any recipe or herbal product that is not approved by the researcher. Long-term treatment (> 2 weeks) with agents that have a high risk of nephrotoxicity or hepatotoxicity unless approved by the medical monitor. Receiving systemic immunosuppressive therapy within 3 months prior to detection.
* Considered by researchers to be unfit to participate in this clinical trial
* Chronic heart failure with ejection fraction less than 30%.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03-30 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-10-30 (Actual)

PRIMARY OUTCOMES:
Adverse effects and Safety | 3 months
  Adverse effects monitoring during and after vaccination

SECONDARY OUTCOMES:
NK transfer Immunogenicity | 6 months
  Measure of NK response against SARS-Cov2 virus

CONTACTS AND LOCATIONS:
Locations (2):
- Colombia (2):
  - Fundacion Salud De Los Andes, Bogotá, Bogotá Distrito Capital
  - Universidad Nacional de Colombia, Bogota, Cundinamarca

IPD SHARING:
Plan to Share IPD: No